CLINICAL TRIAL: NCT03285126
Title: Screening for Eligibility to Participate in a Clinical Trial of Gene Therapy for Late-onset Pompe Disease
Brief Title: Pompe Gene Therapy- Screening for Eligibility
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00085445
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Pompe Disease (Late-onset)
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine eligibility for the future clinical trial of gene therapy in adults with late-onset Pompe disease.

This screening protocol will enroll up to 20 adults patients (>=18 yo) with late-onset Pompe disease. Study assessments include review of medical history, vital signs, physical examination, muscle function testing, lung function testing, blood and urine collection, serum pregnancy test and ECG.

The study results will be collected to perform descriptive statistical analysis and used to determine eligibility for the proposed clinical trial of gene therapy in the future.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Pompe disease by blood or skin fibroblast GAA assay and two pathogenic variants in the GAA gene.
* Age: at least 18 years at enrollment.
* Subjects are capable of giving written consent.
* Receiving ERT at a stable dose for at least 104 weeks.

Exclusion Criteria

* Any condition that would interfere with participation in the study as determined by the principal investigator.
* Pregnancy or nursing mothers.
* History of active hepatitis B, hepatitis C, or cirrhosis
* Receiving any investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with late on-set Pompe Disease.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Eligibility for gene therapy. | Up to 2 days
  The purpose of this study is to determine eligibility for the proposed clinical trial of gene therapy in adults with late-onset Pompe disease. Eligibility is measure by a composite score of blood tests, Electrocardiogram, Pulmonary Function Tests, and Muscle Status Testing.

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Koeberl, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States